CLINICAL TRIAL: NCT04054947
Title: Suicide Prevention in Rural Veterans During High-risk Care Transition Scenarios
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: White River Junction Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Shiner, Staff Psychiatrist, White River Junction Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1439938
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Suicidal and Self-injurious Behavior
Keywords: Suicidal and Self-injurious Behavior
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suicide Prevention Program (Experimental): Behavioral: Suicide Prevention Program Structured care management to improve adherence to discharge planning.
  Interventions: Behavioral: Suicide Prevention Program
- Usual Care (No Intervention): Standard care that occurs as part of mental health treatment

INTERVENTIONS:
Behavioral: Suicide Prevention Program — Structured care management to improve adherence to discharge planning.
  Arms: Suicide Prevention Program

SUMMARY:
In the United States (U.S.), suicide is a major public health concern. U.S. Veterans who live in rural areas may be at even higher risk for suicide than their urban counterparts. Available evidence indicates that suicide risk in rural U.S. Veterans is most concentrated during high-risk care transition scenarios such as discharge from an emergency room. There is limited knowledge about effective interventions to address suicide risk. There is a critical need to develop targeted interventions that address suicide risk during high-risk care transition periods. To be effective, these interventions should address key contributors to suicide risk such as reduced engagement in treatment. This clinical trial evaluates the effect of a suicide prevention intervention to support treatment engagement during high risk transition periods such as discharge from an emergency room.

DETAILED DESCRIPTION:
In the United States (U.S.), death by suicide is a notable public health concern and a particular problem in the U.S. Veteran population. Furthermore, U.S. Veterans who live in rural areas may be at even greater risk for suicide than their urban counterparts. These risks may be concentrated during times of transition in their treatment such as after emergency room discharge. Multiple interventions have been developed to target suicide risk during periods of transition but there is limited evidence regarding their efficacy in preventing suicide. Furthermore, a key contributor to suicide risk may include limited or no engagement in care. Therefore, developing interventions to support engagement in treatment may be effective ways to help mitigate suicide risk and promote participation in care. This clinical trial studies an intervention that is designed to help support treatment engagement during periods of high risk in Veterans who live in rural areas. The trial will recruit Veterans from various treatment settings such as the emergency room, residential drug treatment programs, primary care mental health clinics, and/or inpatient psychiatric units and follow them for a period of six months. The trial evaluates not only the effect of the intervention on suicidal behavior but also measures of engagement.

ELIGIBILITY:
Inclusion Criteria:

Inpatient psychiatric unit:

* Per the unit psychiatrist, hospitalization was due to concerns about acute risk for self-harm including suicidal ideation, suicide attempt, and/or admitting provider deemed the patient was at imminent risk for self-harm
* Be a Veteran eligible to receive VA services
* Be able to speak English

Inpatient medical-surgical unit:

* Received a mental health consultation during admission on the medical-surgical unit
* Per the consult-liaison psychiatrist, patient was recently (within past three months of hospitalization) or is currently at risk for self-harm including suicidal ideation, suicide attempt, or self-harm
* Be a Veteran eligible to receive VA services; be 18 years or older; be able to speak English

Residential Rehabilitation Center (RRC) program:

* Per the RRC treatment team, patient was recently (within past three months of hospitalization) or is currently at risk for self-harm including suicidal ideation, suicide attempt, or self-harm
* Be a Veteran eligible to receive VA services; be 18 years or older; be able to speak English

Primary Mental Health Clinic (PMHC):

* The patient was recently seen for a new evaluation in the WRJ PMHC clinic or a local integrated care clinic that are part of the White River Junction VA Medical Center Catchment Area (i.e., Burlington, Littleton, Rutland, Bennington, Brattleboro, or Keene) by either the mental health nurse practitioner, the psychologist, the psychiatry resident or a psychiatric attending
* The patient is currently at risk for self-harm including suicidal ideation of any severity, suicide attempt, or self-harm; This could have been identified based on a formal suicide assessment scale such as the Columbia Suicide Severity Rating Scale or by clinician assessment as documented in the intake note
* Be a Veteran eligible to receive VA services; be 18 years or older; be able to speak English

Exclusion Criteria:

* Unable to provide informed consent
* Potentially vulnerable populations including prisoners, institutionalized patients, or involuntarily committed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian R Shiner, MD, MPH, Principal Investigator — White River Junction Veterans Affairs Medical Center
Locations (1):
- White River Junction VA Medical Center, White River Junction, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riblet NB, Kenneally L, Stevens S, Watts BV, Gui J, Forehand J, Cornelius S, Rousseau GS, Schwartz JC, Shiner B. A virtual, pilot randomized trial of a brief intervention to prevent suicide in an integrated healthcare setting. Gen Hosp Psychiatry. 2022 Mar-Apr;75:68-74. doi: 10.1016/j.genhosppsych.2022.02.002. Epub 2022 Feb 18. PMID 35202942

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suicide Prevention Program | Usual Care
Started | 31 | 28
Completed | 28 | 23
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Suicide Prevention Program | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.61 (13.73) | 52.97 (15.09) | 51.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 21 | 27 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 30 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 22 | 30 | 52
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 59
The Beck Scale for Suicidal Ideation (BSS) - Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The BSS ranges from 0-38. While there is no established BSS cutoff score to classify suicide risk, there is evidence that higher scores on the BSS correspond to more severe suicidal ideation and that a change of five points or more on the total BSS scores may be clinically relevant. Mean scores at baseline were calculated.
  units on a scale | 9.3 (10.0) | 11.0 (11.1) | 10.2 (10.6)
The Beck Scale for Hopelessness (BHS) - Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The BHS ranges from 0-20 with higher scores associated with increased hopelessness. Mean scores at baseline were calculated.
  units on a scale | 9.7 (6.4) | 9.0 (6.2) | 9.3 (6.3)
The Partners in Health Scale (PIH) (self management) - Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The PIH is used to measure patient self-management of chronic conditions. It is a 12-item instrument, each question measured on a Likert scale of 0-8. Scores range from 0-72. Higher scores indicate better self-management. Mean scores at baseline were calculated.
  units on a scale | 67.2 (12.9) | 67.0 (15.4) | 67.1 (14.2)
The Interpersonal Needs Questionnaire-15: Thwarted Belongingness (INQ-15 TB) -Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The INQ-15 is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item is measured on a 7-point Likert scale, with higher scores suggesting lower perceived connectedness. The score range for the entire scale is 15-105, with the score range for thwarted belongingness being 7-49. Mean scores at baseline were calculated.
  units on a scale | 37.2 (11.0) | 35.4 (14.1) | 36.2 (12.6)
The Interpersonal Needs Questionnaire-15: Perceived Burdensomeness(INQ-15 PB)-Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The INQ-15 is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item is measured on a 7-point Likert scale, with higher scores suggesting lower perceived connectedness. The score range for the entire scale is 15-105, with the score range for perceived burdensomeness being 7-49. The perceived burdensomeness Mean scores at baseline were calculated.
  units on a scale | 17.9 (10.4) | 18.9 (11.2) | 18.5 (10.8)
Multidimensional Scale of Perceived Social Support (MSPSS) - Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — The MSPSS is a 12-item self-reported scale that is designed to ask about support from several sources including friends, family and significant others. The scale has been shown to have good internal and test-retest reliability as well as good validity. The score range is 1-7 with higher values indicating increased perception of social support. Mean scores at baseline were calculated. Population: The MSPSS was added later in the study, after some participants had completed all assessments.
  units on a scale
    number analyzed (Participants) | 19 | 21 | 40
    (all) | 4.4 (1.7) | 4.7 (1.6) | 4.5 (1.6)
Suicide-Related Coping Scale (SRCS) - Mean Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — This scale includes 17 questions related to a patient's perception of their ability to cope with suicidal thoughts. Each item is assessed using a 5-point Likert scale. The scale includes two subscales including an External Coping subscale and an Internal Coping Subscale. The score range for the entire scale is 0-68 with the External Coping being 0-28 and the Internal Coping being 0-28. Higher scores indicate increased perception of suicide-related coping. Mean scores at baseline were calculated. Population: The SRCS was added later in the study, after some participants had completed all assessments.
  units on a scale
    number analyzed (Participants) | 19 | 21 | 40
    (all) | 51.8 (10.4) | 54.5 (10.4) | 53.2 (10.4)

OUTCOME MEASURES:

1. Primary Outcome: The Beck Scale for Suicidal Ideation (BSS)
Description: The BSS ranges from 0-38. While there is no established BSS cutoff score to classify suicide risk, there is evidence that higher scores on the BSS correspond to more severe suicidal ideation and that a change of five points or more on the total BSS scores may be clinically relevant. Mean scores at baseline were calculated.
Time Frame: Change from Baseline BSS at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 28 | 31
score on a scale
  1-month Follow-up: number analyzed (Participants) | 24 | 28
  1-month Follow-up | -2.5 (9.0) | -6.0 (9.9)
  3-month Follow-up: number analyzed (Participants) | 23 | 26
  3-month Follow-up | -2.6 (9.3) | -5.7 (10.1)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | 1.4 (6.5) | -5.3 (8.7)

2. Secondary Outcome: The Beck Scale for Hopelessness (BHS)
Description: The BHS ranges from 0-20 with higher scores associated with increased hopelessness.
Time Frame: Change from Baseline BHS at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 28 | 31
score on a scale
  1-month Follow-up: number analyzed (Participants) | 24 | 28
  1-month Follow-up | -2.1 (5.9) | -3.2 (5.9)
  3-month Follow-up: number analyzed (Participants) | 23 | 26
  3-month Follow-up | -3.0 (6.0) | -4.0 (5.8)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | -0.1 (5.7) | -2.7 (6.0)

3. Secondary Outcome: The Partners in Health Scale (PIH) (Self Management)
Description: The PIH is used to measure patient self-management of chronic conditions. It is a 12-item instrument, each question measured on a Likert scale of 0-8. Scores range from 0-72. Higher scores indicate better self-management. Mean scores at baseline were calculated.
Time Frame: Change from Baseline PIH at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 28 | 31
score on a scale
  1-month Follow-up: number analyzed (Participants) | 24 | 28
  1-month Follow-up | 8.1 (11.7) | 10.4 (14.0)
  3-month Follow-up: number analyzed (Participants) | 23 | 26
  3-month Follow-up | 6.8 (13.0) | 8.1 (14.8)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | 6.2 (12.8) | 4.8 (18.8)

4. Secondary Outcome: The Interpersonal Needs Questionnaire-15: Thwarted Belongingness (INQ-15 TB)
Description: The INQ-15 is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item is measured on a 7-point Likert scale, with higher scores suggesting lower perceived connectedness. The score range for the entire scale is 15-105, with the score range for thwarted belongingness being 7-49. Mean scores at baseline were calculated.
Time Frame: Baseline, 1-month, 3-month, 6-month
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 28 | 31
score on a scale
  1-month Follow-up: number analyzed (Participants) | 24 | 28
  1-month Follow-up | -4.0 (12.2) | -8.2 (13.0)
  3-month Follow-up: number analyzed (Participants) | 23 | 26
  3-month Follow-up | -6.4 (14.0) | -8.7 (13.6)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | 3.4 (15.6) | -5.6 (14.0)

5. Secondary Outcome: Interpersonal Needs Questionnaire 15: Perceived Burdensomeness (INQ-15 PB)
Description: The INQ-15 is a 15-item self-report scale that measures thwarted belongingness (9 items) and perceived burdensomeness (6 items). Each item is measured on a 7-point Likert scale, with higher scores suggesting lower perceived connectedness. The score range for the entire scale is 15-105, with the score range for perceived burdensomeness being 7-49. The perceived burdensomeness Mean scores at baseline were calculated.
Time Frame: Change from Baseline INQ-15 PB at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 28 | 31
score on a scale
  1-month Follow-up: number analyzed (Participants) | 24 | 28
  1-month Follow-up | -1.8 (9.4) | -4.9 (10.0)
  3-month Follow-up: number analyzed (Participants) | 23 | 26
  3-month Follow-up | -4.4 (9.6) | -5.6 (10.4)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | 3.2 (8.3) | -5.9 (10.0)

6. Secondary Outcome: Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a valid and reliable scale that includes a seven-item subscale that asks patients to self-report on actual attempts, interrupted attempts, aborted attempts, and preparatory acts or behaviors.
Time Frame: Number of events according to the CSSR-S at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups.
Measure: Number; unit: number of events
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 28 | 31
number of events
  Baseline | 0 | 0
  1-month Follow-up: number analyzed (Participants) | 24 | 28
  1-month Follow-up | 0 | 0
  3-month Follow-up: number analyzed (Participants) | 23 | 26
  3-month Follow-up | 0 | 0
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | 0 | 0

7. Secondary Outcome: Multidimensional Scale of Perceived Social Support (MSPSS)
Description: The MSPSS is a 12-item self-reported scale that is designed to ask about support from several sources including friends, family and significant others. The scale has been shown to have good internal and test-retest reliability as well as good validity. The score range is 1-7 with higher values indicating increased perception of social support.
Time Frame: Change from Baseline MSPSS at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups. The MSPSS was added later in the study, after some participants had completed all assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 19 | 21
score on a scale
  1-month Follow-up: number analyzed (Participants) | 16 | 18
  1-month Follow-up | 0.6 (1.7) | 0.5 (1.6)
  3-month Follow-up: number analyzed (Participants) | 16 | 16
  3-month Follow-up | 0.7 (1.6) | 1.1 (1.4)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | 0.4 (1.7) | -0.1 (1.9)

8. Secondary Outcome: Suicide-Related Coping Scale (SRCS)
Description: This scale includes 17 questions related to a patient's perception of their ability to cope with suicidal thoughts. Each item is assessed using a 5-point Likert scale. The scale includes two subscales including an External Coping subscale and an Internal Coping Subscale. The score range for the entire scale is 0-68 with the External Coping being 0-28 and the Internal Coping being 0-28. Higher scores indicate increased perception of suicide-related coping. Mean scores at baseline were calculated.
Time Frame: Change from Baseline SRCS at 1-, 3-, and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, 3-, and 6-month follow-ups. The SRCS was added later in the study, after some participants had completed all assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 19 | 21
score on a scale
  1-month Follow-up: number analyzed (Participants) | 16 | 18
  1-month Follow-up | 4.3 (10.4) | 4.7 (9.3)
  3-month Follow-up: number analyzed (Participants) | 16 | 16
  3-month Follow-up | 5.0 (11.0) | 7.9 (9.3)
  6-month Follow-up: number analyzed (Participants) | 6 | 9
  6-month Follow-up | -2.9 (10.5) | 4.4 (12.0)

9. Secondary Outcome: App Engagement Scale (AES) - for Mobile Applications
Description: The App Engagement Scale (AES) is adapted from the end-user version of the Mobile Application Rating Scale (uMARS). The AES has been studied in patients with mental health conditions, has been shown to have good internal reliability, and is strongly related to app engagement. All items are rated on a 5-point scale from "1.Inadequate" to "5.Excellent" with scores ranging from 0 - 40. Higher scores are associated with increased perceived quality of the mobile application.
Time Frame: Change in AES scores at 1- and 6-months
Population: Participants scores were analyzed if they completed the assessment at either baseline, 1-, and 6-month follow-ups. No participants reported using the optional app associated with this study.
Arm/Group | Usual Care | Suicide Prevention Program
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entirety of participant activities (approximately three to six months).
Description: Because our study enrolled a high-risk population, it was expected that patients would potentially report worsening mental health symptoms and/or problems specific to substance use. In some of these cases, these patients would then be expected to be hospitalized or seen in the emergency room to treat these symptoms. Based on local approval from our Institutional Review Board, these events were treated as adverse events.
Arm/Group | Suicide Prevention Program | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 9/31 | 8/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suicide Prevention Program (N=31) | Usual Care (N=28)
Worsening Mental Health (Psychiatric disorders) | 7 (13) | 3 (7) — Events included worsening mental health symptoms. We determined that these adverse events were expected in this high-risk population and unrelated to study procedures.
Alcohol/Substance Use Relapse (Psychiatric disorders) | 3 (4) | 3 (5) — Events included relapse from alcohol and/or other substances. We determined that these adverse events were expected in this high-risk population and unrelated to study procedures.
Cardiac-Related Issues (Cardiac disorders) | 3 (4) | 2 (2) — Events included cardiac-related issues. We determined these adverse events to be unrelated to our study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT04054947/Prot_SAP_002.pdf
  • Informed Consent Form (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT04054947/ICF_001.pdf